CLINICAL TRIAL: NCT04202770
Title: Focused Ultrasound Delivery of Exosomes for Treatment of Refractory Depression, Anxiety, and Neurodegenerative Dementias
Brief Title: Focused Ultrasound and Exosomes to Treat Depression, Anxiety, and Dementias
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending COVID-19 pandemic; pending status of product development
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICSS-2018-018
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Refractory Depression; Anxiety Disorders; Neurodegenerative Diseases
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Anxiety Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: The present study is being undertaken as an open-label study to evaluate the safety and feasibility of exosomes and concurrent focused ultrasound as an intervention for patients with refractory depression, anxiety, and cognitive impairment due to a neurodegenerative disease (e.g., Alzheimer's).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients deemed potentially appropriate candidates for exosome and focused ultrasound therapy for either treatment refractory depression (trMDD), anxiety, or neurodegenerative dementia will be treated with exosomes derived from healthy, full-term Cesarean section amniotic fluid. Up to one hour of transcranial focused ultrasound will be administered immediately prior to exosome treatment in an attempt to facilitate enhanced deployment to the subgenual cingulate for trMDD, the amygdala for anxiety, or the hippocampus for dementia. Target location will be determined by the physician upon enrollment depending on the patient's specific syndrome. Patients will be given 15cc of unconcentrated solution allogenic exosomes (equivalent to 21 million stem cells, Kimera Corporation) intravenously in 200 ccs of normal saline dripped over thirty minutes to one hour.
  Interventions: Other: Exosomes

INTERVENTIONS:
Other: Exosomes — Focused ultrasound delivery of intravenously-infused exosomes

SUMMARY:
This study is designed to evaluate the safety and efficacy of exosome deployment with concurrent transcranial ultrasound in patients with refractory, treatment resistant depression, anxiety, and neurodegenerative dementia.

DETAILED DESCRIPTION:
The present study is designed to enhance the delivery of growth factors and anti-inflammatory agents to localized targets (determined by specific condition) by using focused transcranial ultrasound prior to intravenous infusion of exosomes. Exosomes, which are ubiquitous in blood, body fluids, and tissues are thought to play a normal physiological role in intercellular signaling. Exosomes delivered intravenously can be demonstrated to cross the blood brain barrier naturally. Exosomes and mesenchymal signaling cells (MSC's) demonstrate anti-inflammatory and pro-growth effects in preclinical models and clinical cases reports and have been used intravenously and with intracerebral and intrathecal injection. Various clinical trials have claimed safety and clinical efficacy.

Focused ultrasound has been demonstrated to enhance local blood flow and has been proposed as a non-invasive means of targeting delivery of therapeutic agents. The present paper was designed to use focused ultrasound as a means of enhancing delivery of intravenous exosomes to the subgenual target for patients with refractory depression, the amygdala for patients with anxiety, and the hippocampus for patients with cognitive impairment due to neurodegenerative disease.

ELIGIBILITY:
Inclusion Criteria:

In order for a subject to be considered for the depression application of this study, the following criteria are required:

* Diagnosis of Major Depressive Disorder
* Score greater than 13 on the Beck Depression Inventory
* Failure to remit with 3 antidepressants
* At least 18 years of age

In order for a subject to be considered for the anxiety application of this study, the following criteria are required:

* Diagnosis of Generalized or Acute Anxiety Disorder
* Score greater than 22 on the Beck Anxiety Inventory
* Failure to remit with 3 anxiolytics
* At least 18 years of age

In order for a subject to be considered for the neurodegenerative application of this study, the following criteria are required:

* Cognitive decline with mild cognitive impairment (Clinical Dementia Rating stage 0.5) through moderate dementia (CDR stage 2)
* Lumbar puncture for Abeta 42 and Tau proteins evincing clinical correlation of neurodegenerative disease pathology
* Advanced MRI of the brain including volume measurement of the hippocampus, BOLD, and ASL perfusion scans. On entry, patients will have CDR stage of at least 0.5 and at least one abnormal imaging biomarker. CSF studies have demonstrated good sensitivity and specificity for MCI and dementia of the Alzheimer's type (Tapiola et al., 2009). Additionally, MRI volumetrics and perfusion scans have shown to be useful in differentiating subgroups of AD, PDD/DLB, and FTLD; these values are also responsive to change as patients progress form MCI to dementia (Targosz-Gajniak et al., 2013).

Exclusion Criteria:

* Cognitive decline clearly related to an acute illness
* Subjects unable to give informed consent
* Subjects who would not be able to lay down without excessive movement in a calm environment sufficiently long enough to be able to achieve sleep
* Recent surgery or dental work within 3 months of the scheduled procedure.
* Pregnancy, women who may become pregnant or are breastfeeding
* Advanced terminal illness
* Any active cancer or chemotherapy
* Bone marrow disorder
* Myeloproliferative disorder
* Sickle cell disease
* Primary pulmonary hypertension
* Immunocompromising conditions and/or immunosuppressive therapies
* Any other neoplastic illness or illness characterized by neovascularity
* Macular degeneration
* Subjects with scalp rash or open wounds on the scalp (for example from treatment of squamous cell cancer)
* Advanced kidney, pulmonary, cardiac or liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
[trMDD] Beck Depression Inventory (BDI-II) | 8 weeks from baseline
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
[Anxiety] Beck Anxiety Inventory (BAI) | 8 weeks from baseline
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
[Dementia] Quick Dementia Rating Scale (QDRS) | 8 weeks from baseline
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).
[ALL] Global Rating of Change (GRC) | 8 weeks from baseline
  The GRC consists of a single likert-scale ranging from "-5" (very much worse) to "0" (neutral/no change) to "5" (very much better). The GRC is obtained in an interview format to assess a patient's perceived change in status following a treatment. A score that is at least 2 or greater is considered to indicate clinically significant change.

SECONDARY OUTCOMES:
[trMDD] Patient Depression Questionnaire (PDQ-9) | 8 weeks from baseline
  The PDQ-9 is a 9-item, self-report questionnaire to evaluate for depressive symptoms. Each question asks the patient if they have experienced a particular depressive symptom over the past two weeks. Answers may range from "0" (not at all), "1" (several days/week), "2" (more than half of the days), and "3" (nearly every day). Maximum total score is 27 points. A higher score indicates more severe depressive symptoms. A reduction in total score by at least 30% is considered clinically meaningful.
[trMDD] Hamilton Depression Rating Scale (HAM-D) | 8 weeks from baseline
  The HAM-D is a 17-item, interview style questionnaire. A trained staff member administers this form to a patient and scores the patients' responses on a scale of "0" (symptom absent) to "4" (most severe option per symptom). A higher total score indicates a more severe level of depression. The maximum possible score is 50 points. A change in score of at least 30% is considered clinically meaningful.
[Anxiety] Hamilton Anxiety Rating Scale (HAM-A) | 8 weeks from baseline
  The HAM-A is an observer/rater scale consisting of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
[Dementia] Repeatable Battery Assessment of Neuropsychological Status (RBANS) versions A-D | 8 weeks from baseline
  RBANS assesses immediate memory, visuospatial skill, language, attention, and delayed memory. Patient performance on each subscale immediate memory, language, attention, visuospatial, and delayed memory are scored relative to validated norms for same-aged peers. A change of 8+ points in the Total Scale score, 11+ points in the Immediate Memory score, 9+ points in the Language score, 4+ points on the Attention score, 14+ points is considered significant for the Visuospatial score, and 10+ points for the Delayed Memory score are considered significant.
[Dementia] Montreal Cognitive Assessment (MoCA) versions 7.1-7.3 | 8 weeks from baseline
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, M.D., Principal Investigator — Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West Los Angeles, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be made publicly available due to ethical and privacy concerns. Anonymized data will be available upon reasonable request from any qualified investigator.

REFERENCES:
- [Background] Bandelow B, Michaelis S. Epidemiology of anxiety disorders in the 21st century. Dialogues Clin Neurosci. 2015 Sep;17(3):327-35. doi: 10.31887/DCNS.2015.17.3/bbandelow. PMID 26487813
- [Background] Coupe P, Manjon JV, Lanuza E, Catheline G. Lifespan Changes of the Human Brain In Alzheimer's Disease. Sci Rep. 2019 Mar 8;9(1):3998. doi: 10.1038/s41598-019-39809-8. PMID 30850617
- [Background] Ferrari AJ, Charlson FJ, Norman RE, Patten SB, Freedman G, Murray CJ, Vos T, Whiteford HA. Burden of depressive disorders by country, sex, age, and year: findings from the global burden of disease study 2010. PLoS Med. 2013 Nov;10(11):e1001547. doi: 10.1371/journal.pmed.1001547. Epub 2013 Nov 5. PMID 24223526
- [Background] Hebron ML, Lonskaya I, Moussa CE. Nilotinib reverses loss of dopamine neurons and improves motor behavior via autophagic degradation of alpha-synuclein in Parkinson's disease models. Hum Mol Genet. 2013 Aug 15;22(16):3315-28. doi: 10.1093/hmg/ddt192. Epub 2013 May 10. PMID 23666528
- [Background] Pagan, F., Valadez, E., Torres-Yaghi, Y., Falconer, R., Mills, R., Rogers, S., Wilmarth, B., Hebron, M., & Moussa, C. (2016) Effects of nilotinib on safety in open-label phase I clinical trial in Parkinson's disease with dementia and Lewy body dementia. Movement Disorders, 31(2).
- [Background] Montgomery SA, Baldwin DS, Riley A. Antidepressant medications: a review of the evidence for drug-induced sexual dysfunction. J Affect Disord. 2002 May;69(1-3):119-40. doi: 10.1016/s0165-0327(01)00313-5. PMID 12103459
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Cipriani A, Furukawa TA, Salanti G, Geddes JR, Higgins JP, Churchill R, Watanabe N, Nakagawa A, Omori IM, McGuire H, Tansella M, Barbui C. Comparative efficacy and acceptability of 12 new-generation antidepressants: a multiple-treatments meta-analysis. Lancet. 2009 Feb 28;373(9665):746-58. doi: 10.1016/S0140-6736(09)60046-5. PMID 19185342
- [Background] Setiawan E, Attwells S, Wilson AA, Mizrahi R, Rusjan PM, Miler L, Xu C, Sharma S, Kish S, Houle S, Meyer JH. Association of translocator protein total distribution volume with duration of untreated major depressive disorder: a cross-sectional study. Lancet Psychiatry. 2018 Apr;5(4):339-347. doi: 10.1016/S2215-0366(18)30048-8. Epub 2018 Feb 26. PMID 29496589
- [Background] Drevets WC, Savitz J, Trimble M. The subgenual anterior cingulate cortex in mood disorders. CNS Spectr. 2008 Aug;13(8):663-81. doi: 10.1017/s1092852900013754. PMID 18704022
- [Background] Lozano AM, Mayberg HS, Giacobbe P, Hamani C, Craddock RC, Kennedy SH. Subcallosal cingulate gyrus deep brain stimulation for treatment-resistant depression. Biol Psychiatry. 2008 Sep 15;64(6):461-7. doi: 10.1016/j.biopsych.2008.05.034. Epub 2008 Jul 18. PMID 18639234
- [Background] Jalbrzikowski M, Larsen B, Hallquist MN, Foran W, Calabro F, Luna B. Development of White Matter Microstructure and Intrinsic Functional Connectivity Between the Amygdala and Ventromedial Prefrontal Cortex: Associations With Anxiety and Depression. Biol Psychiatry. 2017 Oct 1;82(7):511-521. doi: 10.1016/j.biopsych.2017.01.008. Epub 2017 Jan 17. PMID 28274468
- [Background] Mayberg H. Depression, II: localization of pathophysiology. Am J Psychiatry. 2002 Dec;159(12):1979. doi: 10.1176/appi.ajp.159.12.1979. No abstract available. PMID 12450943
- [Background] Mayberg HS. Limbic-cortical dysregulation: a proposed model of depression. J Neuropsychiatry Clin Neurosci. 1997 Summer;9(3):471-81. doi: 10.1176/jnp.9.3.471. PMID 9276848
- [Background] Mayberg HS. Modulating limbic-cortical circuits in depression: targets of antidepressant treatments. Semin Clin Neuropsychiatry. 2002 Oct;7(4):255-68. doi: 10.1053/scnp.2002.35223. PMID 12382208
- [Background] Mayberg HS. Modulating dysfunctional limbic-cortical circuits in depression: towards development of brain-based algorithms for diagnosis and optimised treatment. Br Med Bull. 2003;65:193-207. doi: 10.1093/bmb/65.1.193. PMID 12697626
- [Background] Mayberg HS. Positron emission tomography imaging in depression: a neural systems perspective. Neuroimaging Clin N Am. 2003 Nov;13(4):805-15. doi: 10.1016/s1052-5149(03)00104-7. PMID 15024963
- [Background] Mayberg HS. Defining the neural circuitry of depression: toward a new nosology with therapeutic implications. Biol Psychiatry. 2007 Mar 15;61(6):729-30. doi: 10.1016/j.biopsych.2007.01.013. No abstract available. PMID 17338903
- [Background] Mayberg HS. Targeted electrode-based modulation of neural circuits for depression. J Clin Invest. 2009 Apr;119(4):717-25. doi: 10.1172/JCI38454. PMID 19339763
- [Background] Mayberg HS, Brannan SK, Mahurin RK, Jerabek PA, Brickman JS, Tekell JL, Silva JA, McGinnis S, Glass TG, Martin CC, Fox PT. Cingulate function in depression: a potential predictor of treatment response. Neuroreport. 1997 Mar 3;8(4):1057-61. doi: 10.1097/00001756-199703030-00048. PMID 9141092
- [Background] Mayberg HS, Liotti M, Brannan SK, McGinnis S, Mahurin RK, Jerabek PA, Silva JA, Tekell JL, Martin CC, Lancaster JL, Fox PT. Reciprocal limbic-cortical function and negative mood: converging PET findings in depression and normal sadness. Am J Psychiatry. 1999 May;156(5):675-82. doi: 10.1176/ajp.156.5.675. PMID 10327898
- [Background] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841
- [Background] Botteron KN, Raichle ME, Drevets WC, Heath AC, Todd RD. Volumetric reduction in left subgenual prefrontal cortex in early onset depression. Biol Psychiatry. 2002 Feb 15;51(4):342-4. doi: 10.1016/s0006-3223(01)01280-x. PMID 11958786
- [Background] Yucel K, McKinnon M, Chahal R, Taylor V, Macdonald K, Joffe R, Macqueen G. Increased subgenual prefrontal cortex size in remitted patients with major depressive disorder. Psychiatry Res. 2009 Jul 15;173(1):71-6. doi: 10.1016/j.pscychresns.2008.07.013. Epub 2009 May 21. PMID 19464154
- [Background] Riva-Posse P, Choi KS, Holtzheimer PE, Crowell AL, Garlow SJ, Rajendra JK, McIntyre CC, Gross RE, Mayberg HS. A connectomic approach for subcallosal cingulate deep brain stimulation surgery: prospective targeting in treatment-resistant depression. Mol Psychiatry. 2018 Apr;23(4):843-849. doi: 10.1038/mp.2017.59. Epub 2017 Apr 11. PMID 28397839
- [Background] Yuan D, Zhao Y, Banks WA, Bullock KM, Haney M, Batrakova E, Kabanov AV. Macrophage exosomes as natural nanocarriers for protein delivery to inflamed brain. Biomaterials. 2017 Oct;142:1-12. doi: 10.1016/j.biomaterials.2017.07.011. Epub 2017 Jul 10. PMID 28715655
- [Background] Boshuizen MCS, Steinberg GK. Stem Cell-Based Immunomodulation After Stroke: Effects on Brain Repair Processes. Stroke. 2018 Jun;49(6):1563-1570. doi: 10.1161/STROKEAHA.117.020465. Epub 2018 May 3. No abstract available. PMID 29724892
- [Background] Detante O, Rome C, Papassin J. How to use stem cells for repair in stroke patients. Rev Neurol (Paris). 2017 Nov;173(9):572-576. doi: 10.1016/j.neurol.2017.09.003. Epub 2017 Oct 21. PMID 29033030
- [Background] Doeppner TR, Bahr M, Hermann DM, Giebel B. Concise Review: Extracellular Vesicles Overcoming Limitations of Cell Therapies in Ischemic Stroke. Stem Cells Transl Med. 2017 Nov;6(11):2044-2052. doi: 10.1002/sctm.17-0081. Epub 2017 Sep 23. PMID 28941317
- [Background] Sarmah D, Agrawal V, Rane P, Bhute S, Watanabe M, Kalia K, Ghosh Z, Dave KR, Yavagal DR, Bhattacharya P. Mesenchymal Stem Cell Therapy in Ischemic Stroke: A Meta-analysis of Preclinical Studies. Clin Pharmacol Ther. 2018 Jun;103(6):990-998. doi: 10.1002/cpt.927. Epub 2017 Dec 14. PMID 29090465
- [Background] Stonesifer C, Corey S, Ghanekar S, Diamandis Z, Acosta SA, Borlongan CV. Stem cell therapy for abrogating stroke-induced neuroinflammation and relevant secondary cell death mechanisms. Prog Neurobiol. 2017 Nov;158:94-131. doi: 10.1016/j.pneurobio.2017.07.004. Epub 2017 Jul 23. PMID 28743464
- [Background] Sussman ES, Steinberg GK. A Focused Review of Clinical and Preclinical Studies of Cell-Based Therapies in Stroke. Neurosurgery. 2017 Sep 1;64(CN_suppl_1):92-96. doi: 10.1093/neuros/nyx329. No abstract available. PMID 28899062
- [Background] Suzuki E, Fujita D, Takahashi M, Oba S, Nishimatsu H. Therapeutic Effects of Mesenchymal Stem Cell-Derived Exosomes in Cardiovascular Disease. Adv Exp Med Biol. 2017;998:179-185. doi: 10.1007/978-981-10-4397-0_12. PMID 28936740
- [Background] Tapiola T, Alafuzoff I, Herukka SK, Parkkinen L, Hartikainen P, Soininen H, Pirttila T. Cerebrospinal fluid beta-amyloid 42 and tau proteins as biomarkers of Alzheimer-type pathologic changes in the brain. Arch Neurol. 2009 Mar;66(3):382-9. doi: 10.1001/archneurol.2008.596. PMID 19273758
- [Background] Targosz-Gajniak MG, Siuda JS, Wicher MM, Banasik TJ, Bujak MA, Augusciak-Duma AM, Opala G. Magnetic resonance spectroscopy as a predictor of conversion of mild cognitive impairment to dementia. J Neurol Sci. 2013 Dec 15;335(1-2):58-63. doi: 10.1016/j.jns.2013.08.023. Epub 2013 Aug 27. PMID 24035276
- [Background] Toyoshima A, Yasuhara T, Date I. Mesenchymal Stem Cell Therapy for Ischemic Stroke. Acta Med Okayama. 2017 Aug;71(4):263-268. doi: 10.18926/AMO/55302. PMID 28824181
- [Background] Mah L, Szabuniewicz C, Fiocco AJ. Can anxiety damage the brain? Curr Opin Psychiatry. 2016 Jan;29(1):56-63. doi: 10.1097/YCO.0000000000000223. PMID 26651008
- [Background] McDannold N, Vykhodtseva N, Hynynen K. Blood-brain barrier disruption induced by focused ultrasound and circulating preformed microbubbles appears to be characterized by the mechanical index. Ultrasound Med Biol. 2008 May;34(5):834-40. doi: 10.1016/j.ultrasmedbio.2007.10.016. Epub 2008 Jan 22. PMID 18207311